CLINICAL TRIAL: NCT05913271
Title: Study on the Correlation Between NAT2(N-acetyltransferase2) Gene Polymorphism and CrCl(Creatine Clreance) and the Efficacy and Safety of Levosimendan in Patients With Severe Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yi Han (Other)
Collaborators: Qianfoshan Hospital (Other)
Responsible Party: Sponsor-Investigator, Yi Han, Associate professor of pharmacy, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: LNAT
Record Dates: First submitted 2023-06-08; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure; Levosimendan; Efficacy; Safety
Keywords: Severe Heart Failure; Levosimendan; NAT2(N-acetyltransferase2) Gene Polymorphism; CrCl(Creatine clreance)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 35 Days
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To evaluate the efficacy and safety of levosimendan in the treatment of heart failure ;
2. Guide patients to apply levosimendan individually and establish a dose adjustment program.

DETAILED DESCRIPTION:
The efficacy and safety of levosimendan in Chinese patients with different acetylmetabolites and CrCl(Creatine clreance) were re-evaluated after marketing. The population pharmacokinetics of different populations was studied, and the patients were guided to apply levosimendan individually and establish a dose adjustment program.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Patients who were clearly diagnosed with heart failure ( cardiac insufficiency ) and LVEF(Left Ventricular Ejection Fraction) < 50 %, and were judged by the physician to need and agree to use levosimendan to maintain hemodynamic stability
* Sign informed consent

Exclusion Criteria:

* chronic heart failure and New York Heart Association ( NYHA ) class I ~ II
* Complicated with infective endocarditis, aortic dissection, severe liver dysfunction ( child-pugh C ), severe renal insufficiency ( CrCl < 30 ml / min ), hypertrophic obstructive cardiomyopathy, ventricular assist device or surgical cardiac surgery within 30 days before the use of levosimendan
* Patients with severe ventricular arrhythmia 1 within 24 hours before levosimendan and systolic blood pressure 100 times / min within 2 hours before levosimendan
* During hospitalization, other positive inotropic drugs 2 were used when levosimendan was intravenously pumped or dripped, excluding the use of catecholamines for rescue
* received positive inotropic drug 2 treatment in the last 30 days
* Lack of serum creatinine, brain natriuretic peptide or brain natriuretic peptide precursor, serum total bilirubin, cardiac ultrasound baseline ( within 14 days before using levosimendan ) data
* pregnant and lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe heart failure generally refers to the low perfusion of tissues and organs caused by acute heart failure and acute exacerbation of chronic cardiac insufficiency, which seriously affects life. It is often combined with multiple organs, especially renal function injury. Its prognosis is poor, mortality and readmission rate are high, and the 1-year mortality rate can reach more than 20 %.
Sampling Method: Non-Probability Sample
Enrollment: 352 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
35-day survival rate | 35-day
  Survival of patients at 35 days

SECONDARY OUTCOMES:
The changes of plasma BNP(brain natriuretic peptide） / NT-proBNP（N-terminal B-type natriuretic peptide） before and after treatment. | 35-day
  Measurement of BNP（brain natriuretic peptide） / NT-proBNP（N-terminal B-type natriuretic peptide）
The improvement rate of patients ' health status | 35-day
  EQ-5D scale(EuroQol Five Dimensions Questionnaire) was used to assess health status
The incidence of composite endpoint events ( within 35 days ) included mortality, unplanned readmission, transfer to ICU, and rescue. | 35-day
  Incidence of composite endpoint events within 35 days

OTHER OUTCOMES:
The incidence of adverse reactions, including headache, hypotension, arrhythmia. | 35-day
  Adverse reactions after medication

CONTACTS AND LOCATIONS:
Overall Officials: Yi Han, doctorate, Principal Investigator — First Affiliated Hospital of Shandong First Medical University ( Qianfoshan Hospital of Shandong Province )
Locations (1):
- First Affiliated Hospital of Shandong First Medical University ( Qianfoshan Hospital of Shandong Province ), Jinan, Shandong, China